CLINICAL TRIAL: NCT06968520
Title: Correlation and Predictive Study of Metal Elements in Radiation-Induced Oral Mucositis: A Prospective, Longitudinal Cohort Study
Brief Title: Correlation and Predictive Research of Metal Elements in Radiation-Induced Oral Mucositis
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NEFC-2025-173
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Tumors; Metal; Copper; Radiotherapy-Induced Oral Mucositis
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiotherapy is the main treatment method for head and neck tumors. However, almost all patients with head and neck tumors will develop acute inflammatory reactions such as Radiotherapy-Induced Oral Mucositis (RIOM) after receiving Radiotherapy, resulting in a decline in the quality of life of patients, hindering the smooth implementation of the treatment plan, reducing the therapeutic effect, and increasing the economic burden of patients. However, the current treatment strategies for RIOM focus on symptomatic treatment and have little impact on the course, severity and related complications of mucositis. Therefore, exploring effective strategies, predicting the incidence and severity of RIOM in patients, and providing prevention and treatment are the clinical bottlenecks and cutting-edge issues that urgently need to be solved in the current clinical practice of radiotherapy for head and neck tumors. Previous studies have shown that the steady-state of metallic elements may be closely related to the occurrence and development of RIOM. Therefore, we plan to conduct a prospective, single-center, observational study to further explore the correlation between metal elements and severe RIOM, analyze its predictive efficacy, and observe the dynamic changes of metal elements in radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1）Sign the informed consent form; 2) Confirmed by pathological biopsy as nasopharyngeal carcinoma or head and neck tumors; 3) Have indications for radiotherapy and voluntarily accept radiotherapy; 4) ECOG PS: 0/1; 5) Age: 18-75 years old; 6) Laboratory tests confirm good organ function.

Exclusion Criteria:

1. There are contraindications for radiotherapy;
2. Combined with other tumors;
3. Pathological sections could not be obtained;
4. The patient has any serious concurrent diseases that may pose unacceptable risks or have a negative impact on trial compliance. For instance, unstable heart diseases requiring treatment, chronic hepatitis, kidney diseases with poor conditions, uncontrolled diabetes (fasting blood glucose greater than 1.5 × ULN), and mental disorders;
5. The researcher judged that it was not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the 2021CSCO guidelines, patients diagnosed as nasopharyngeal carcinoma and head and neck tumors were standardized
Sampling Method: Non-Probability Sample
Enrollment: 383 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The incidence rates of severe radiation-induced oral mucositis. | Through study completion, up to 1 year
  The incidence rates of sever radiation-induced oral mucositis across various severity grades will be determined.Grade>=3 is regarded as severe RTOM.

SECONDARY OUTCOMES:
Duration of RTOM and SRTOM. | Through study completion, up to 1 year
  Recording the start time and duration of RTOM and SRTOM.
Quality of life score. | Through study completion, up to 1 year
  The quality of life including physical health, mental health, spiritual health and social and interpersonal relationships.
Other recent adverse radiation reactions | Through study completion, up to 1 year
  Other recent adverse radiation reactions caused by radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang hospital, Southern medical university, Guangzhou, Guangdong, China